CLINICAL TRIAL: NCT05710107
Title: The Impact or Quadratum Lumborum (QL) Block Versus Pericapsular Nerve Group (PENG) With Lateral Femoral Cutaneous (LFC) Nerve Blocks for Analgesia After Hip Arthroplasty: a Prospective, Randomized Clinical Trial
Brief Title: QL vs PENG for Analgesia After Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Ellen Hay, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Pro00124880
Record Dates: First submitted 2023-01-12; First posted 2023-02-02 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Block; Hip Replacement; Postoperative Pain
MeSH Terms: conditions — Bites and Stings; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Subjects, surgeons, and data collectors will all be blinded to the allocated group. Unblinded personnel will be the Anesthesia Attending placing the block and clinical staff assisting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PENG + LFC Block (Active Comparator): The pericapsular nerve group (PENG) block is an ultrasound-guided approach, first described by Giron-Arango et al. for the blockade of the articular branches of the femoral, obturator and accessory obturator nerves that provide sensory innervation to the anterior hip capsule [5,6]. In the PENG block, a low-frequency, curvilinear probe is used to visualize the anterior inferior iliac spine, iliopsoas tendon, and iliopubic eminence. After placing a subcutaneous skin wheel with lidocaine, a blunt regional anesthesia needle is inserted using in-plane ultrasound guidance. The needle is advanced until the tip lies on the lateral and inferior margin of the iliopsoas tendon between the anterior inferior iliac spine (lateral) and iliopubic eminence (deep).
  Interventions: Other: PENG + LFC Block
- QL Block (Active Comparator): The lateral QL block is performed by injecting local anesthetic deep to the transversus abdominis aponeurosis and superficial to the fascia transversalis with direct ultrasound guidance. After completing consent, placing monitors and providing mild sedation, the patient is positioned laterally and the muscular anatomy (external oblique, internal oblique, transverse abdominis, quadratus lumborum and latissimus dorsi muscles) identified. After placing a subcutaneous skin wheel with lidocaine, a blunt regional anesthesia needle is inserted using in-plane ultrasound guidance. Local anesthetic is deposited incrementally with frequent aspiration in the anterolateral border of the quadratus lumborum muscle at the junction of the transversalis fascia, outside the anterior layer of the thoracolumbar fascia and superficial to the fascia transversalis.
  Interventions: Other: QL Block

INTERVENTIONS:
Other: PENG + LFC Block — Subjects assigned to this group will receive PENG + LFC Block
  Arms: PENG + LFC Block
Other: QL Block — Subjects randomized to this group will receive a QL Block
  Arms: QL Block

SUMMARY:
This study will consist of patients 18 years and older who are undergoing elective hip replacement with planned same day discharge. The patients will be randomized to receive a PENG+LFC or QL block prior to undergoing the surgery to help with postoperative pain control. The primary goal will be assessing postoperative opioid use during the first 72 hours after surgery. Secondary outcomes will include postoperative pain scores from, 0-72 hours. Additional outcomes consist of time to first ambulation, functional and mobility outcomes, PACU duration, patient satisfaction and opioid related side effects.

DETAILED DESCRIPTION:
1. Patients demographic data and health information will be collected including age, height, weight, and details related to injury from the medical record. Patients will also be asked to complete a set of questionnaires detailing how they feel prior to the procedure.
2. Patients will be randomly assigned to one of two groups. Group A will receive the PENG + LFC block. Group B will receive the QL block. Patients will be sedated while receiving either block.

   If patients are assigned to the QL block, ultrasound technology will be used to identify appropriate structures on the side of the abdomen. An injection of lidocaine (numbing medication) into the skin will be inserted first for comfort. A second needle will be inserted into the side of the abdomen and a numbing medication called ropivacaine will be injected.\

   If patients are randomized to receive PENG + LFC, ultrasound technology will be used to identify appropriate structures between the hip and groin area. An injection of lidocaine (numbing medication) into the skin will be inserted first for comfort. A needle will be inserted to the appropriate location between the hip and groin, and a numbing medication called ropivacaine will be injected. This may take more than one injection in the same area.
3. Surgery will begin shortly after the placement of the nerve block(s).
4. Before being discharged from the surgery center, patients will be asked their current pain score (0-100) and the study team will provide a detailed information sheet that includes instructions for the study follow-up period. Patients will receive a text message with a link to a questionnaire at 9:00 AM, and 3:00 PM for the first three days after surgery. This questionnaire will ask them to rate their average pain at rest and while moving in a specific time period by using a visual scale from 0-100. The study will also ask questions about the pain medication taken in that same time period. At day 7, participants will receive a survey link via text message with additional questions about recovery. If they do not wish to be contacted by text message, someone from the study team will contact them by telephone at the end of the seven days and ask them to read back the information recorded on the paper data sheet provided.
5. At approximately 2-3 weeks after surgery, and again at approximately 6 weeks after surgery a study team member will contact patients either via telephone or visit patients during their post-surgical clinic visit to complete a set of questionnaires related to their recovery. Patients will also be asked to report any side effects, urgent care/emergency room visits, or any new conditions while participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 18 years of age
* undergoing elective hip arthroplasty with planned same day discharge

Exclusion Criteria:

* local anesthetic allergy
* subjects with a weight less than 40kg
* subjects that are unable or choose not to give informed consent
* Known preoperative substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-11-12 (Actual); Study Completion 2023-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Hay, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hay E, Kelly T, Wolf BJ, Hansen E, Brown A, Lautenschlager C, Wilson SH. Comparison of pericapsular nerve group and lateral quadratus lumborum blocks on cumulative opioid consumption after primary total hip arthroplasty: a randomized controlled trial. Reg Anesth Pain Med. 2024 Oct 10:rapm-2024-105875. doi: 10.1136/rapm-2024-105875. Online ahead of print. PMID 39389587

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PENG + LFC Block | QL Block
Started | 53 | 53
Completed (53 subjects began the study. in the PENG + LFC group 3 subjects were removed and their data was not included (1 subject withdrew, and 2 were unable to have the assigned block performed) bringing the total to 50. 53 subjects began in the QL block group and 2 were removed (1 voluntarily withdrew and 1 was withdrawn by the study team) bringing the total to 51 included in this group. Lost to follow up were included in analysis but had missing data.) | 42 | 42
Not Completed | 11 | 11
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 8 | 9
Not completed — Unable to place assigned block | 2 | 0
Not completed — Withdrawn by study team | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PENG + LFC Block | QL Block | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (12.7) | 65.8 (9.77) | 64.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 29 | 51
  Male | 28 | 22 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 34 | 42 | 76
  Black, African American, or Other | 16 | 9 | 25
Average hip pain with movement in the last week [Mean (Standard Deviation); unit: units on a scale] — Before surgery, participants were asked to rate their average hip pain with movement in the past week using a Visual Analog Scale (VAS) from 0-100. A higher number means worse pain.
  units on a scale | 67.1 (23.7) | 66.7 (18.9) | 66.9 (21.3)
Average hip pain at rest in the last week [Mean (Standard Deviation); unit: units on a scale] — Before surgery, participants were asked to rate their average hip pain while at rest in the past week using a Visual Analog Scale (VAS) from 0-100. A higher number means worse pain.
  units on a scale | 43.9 (30.3) | 44.3 (25.4) | 44.1 (27.8)

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Cumulative Opioid Consumption
Description: The primary outcome will be postoperative cumulative opioid consumption (in IV morphine mg equivalents: IV MME) over time, from 0-72 hours postoperatively. Cumulative opioid consumption will be evaluated at PACU, and through 72 hours post-op.
Time Frame: 0-72 hours postoperatively
Measure: Mean (95% Confidence Interval); unit: morphine milligram equivalents
Arm/Group | PENG + LFC Block | QL Block
Number analyzed (Participants) | 50 | 51
morphine milligram equivalents
  PACU | 12.7 [0.0 to 29.8] | 9.9 [0.0 to 26.8]
  PACU through 12-hours post-op | 29.4 [12.8 to 46.0] | 23.2 [6.8 to 39.6]
  PACU through 24-hours post-op | 46.1 [29.6 to 62.6] | 36.4 [20.2 to 52.6]
  PACU through 36-hours post op | 62.8 [46.1 to 79.5] | 49.7 [33.4 to 66.0]
  PACU through 48-hours post-op | 79.5 [62.2 to 96.8] | 63.0 [46.3 to 79.7]
  PACU through 60-hours post-op | 96.2 [78.0 to 114.5] | 76.3 [58.8 to 93.7]
  PACU to 72-hours post-op | 112.9 [93.4 to 132.4] | 89.5 [71.1 to 107.9]

2. Secondary Outcome: Average Postoperative Pain Score
Description: Average postoperative pain score on the visual analog scale (VAS) from 0-100 from 0-72-hours post-op, including approximately 60 minutes after PACU arrival. The lower the reported pain score, the better the outcome.
Time Frame: 0-72 hours postoperatively
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PENG + LFC Block | QL Block
Number analyzed (Participants) | 50 | 51
units on a scale
  60 minutes after PACU Arrival | 33.2 [26.5 to 39.9] | 29.5 [22.9 to 36.1]
  12-hours post-op | 47.2 [39.2 to 55.1] | 43.5 [36.5 to 50.6]
  24-hours post-op | 48.7 [40.5 to 60.8] | 45.1 [38.7 to 51.5]
  36-hours post-op | 46.0 [38.3 to 53.8] | 42.4 [35.7 to 49.1]
  48-hours post-op | 40.4 [32.4 to 48.4] | 36.8 [29.8 to 43.8]
  60-hours post-op | 38.3 [29.5 to 47.2] | 34.7 [27.9 to 41.5]
  72-hours post-op | 35.3 [27.1 to 43.5] | 31.7 [24.8 to 38.6]

3. Other Pre Specified Outcome: Time to First Ambulation
Description: How many minutes after anesthesia stop time patients first ambulate
Time Frame: From anesthesia stop time to first ambulation in minutes, assessed up to 7 days post-op.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | PENG + LFC Block | QL Block
Number analyzed (Participants) | 50 | 51
minutes | 500.5 [217 to 3031] | 502 [204 to 1628]

4. Other Pre Specified Outcome: PROMIS Physical Health
Description: The PROMIS (Patient-Reported Outcomes Measurement Information System) Global Health Questionnaire assesses functional outcomes such by evaluating the patient's physical aspects of health using the subscale, PROMIS Physical Health, at 1 week post-op, 2 weeks post-op, and 6 weeks post-op. The physical health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score between 16.2-67.7. The population mean is 50 and SD is 10. Higher T scores represent better physical health. Values are reported as constructed T scores.
Time Frame: Up to 6 weeks post-operatively
Measure: Mean (95% Confidence Interval); unit: T scores
Arm/Group | PENG + LFC Block | QL Block
Number analyzed (Participants) | 50 | 51
T scores
  1 Week Post-Op | 42.6 [40.4 to 44.9] | 43.0 [40.7 to 45.2]
  2 Weeks Post-Op | 46.0 [43.8 to 48.3] | 46.4 [44.1 to 48.7]
  6 Weeks Post-Op | 48.0 [45.7 to 50.2] | 48.3 [46.1 to 50.5]

5. Other Pre Specified Outcome: Overall Hip Health
Description: The HOOS Jr will assess overall Hip Health in participants at 1 week post-op, 2 weeks post-op, and 6 weeks post-op. HOOS-JR is scored by summing the raw response (range 0-24) and then converting it to an interval score using a table provided. The interval score ranges from 0 to 100 where 0 represents total hip disability and 100 represents perfect hip health.
Time Frame: Up to 6 weeks post-operatively
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PENG + LFC Block | QL Block
Number analyzed (Participants) | 50 | 51
units on a scale
  1 week post-op | 54.3 [49.2 to 59.4] | 57.2 [53.0 to 61.4]
  2 weeks post-op | 62.3 [58.1 to 66.6] | 65.3 [60.8 to 69.8]
  6 weeks post-op | 68.9 [64.9 to 72.9] | 71.8 [67.3 to 76.3]

6. Other Pre Specified Outcome: PACU Duration
Description: Time patient spent in PACU defined as surgery end time, to the time discharged from PACU.
Time Frame: surgery end to time discharged from PACU, assessed up to 6 weeks post-op
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | PENG + LFC Block | QL Block
Number analyzed (Participants) | 50 | 51
minutes | 295 [29 to 553] | 293 [34 to 547]

7. Other Pre Specified Outcome: PROMIS Mental Health
Description: The PROMIS (Patient-Reported Outcomes Measurement Information System) Mental Health Questionnaire will assess functional outcomes such by evaluating the patient's physical aspects of health using the subscale, PROMIS Physical Health, at 1 week post-op, 2 weeks post-op, and 6 weeks post-op. The physical health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score between 21.2-67.6. The population mean is 50 and SD is 10. Higher T scores represent better mental health. Values are reported as constructed T scores.
Time Frame: up to 6 weeks post-operatively
Measure: Mean (95% Confidence Interval); unit: T scores
Arm/Group | PENG + LFC Block | QL Block
Number analyzed (Participants) | 50 | 51
T scores
  1 week post-op | 45.9 [43.9 to 47.9] | 46.2 [44.2 to 48.3]
  2 weeks post-op | 49.0 [47.0 to 60.0] | 49.3 [47.3 to 51.3]
  6 weeks post-op | 50.7 [48.7 to 52.8] | 51.0 [49.1 to 52.9]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time the participant signed the consent document and was randomized, to 6 weeks post-op.
Arm/Group | PENG + LFC Block | QL Block
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 30/50 | 28/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PENG + LFC Block (N=50) | QL Block (N=51)
Itching (Skin and subcutaneous tissue disorders) | 19 (19) | 22 (22)
Nausea (Gastrointestinal disorders) | 14 (14) | 9 (9)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Leg Swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prolonged numbness from spinal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional Numbness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rash, shingles (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Post-Operative Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower extremity sensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT05710107/Prot_SAP_000.pdf